CLINICAL TRIAL: NCT04049708
Title: Intrarater Reliability in Different Days and Interrater Reliability of Physical Function Assessment in HD Patients
Brief Title: Intrarater and Interrater Reliability Physical Function Measures in HD BCN
Acronym: ReliabilityBCN
Status: Completed | Type: Observational
Sponsor: Cardenal Herrera University (Other)
Collaborators: Consorci Sanitari de Terrassa. Hospital de Terrassa (Unknown)
Responsible Party: Principal Investigator, Eva Segura Ortí, Professor, Cardenal Herrera University
Other Study IDs: ReliabilityBCN
Record Dates: First submitted 2019-08-05; First posted 2019-08-08 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: End Stage Renal Disease on Dialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Reliability of physical function — Test-retest reliability of physical function in hemodialysis patients

SUMMARY:
The investigators will calculate values of absolute and relative reliability for intrarater reliability when the measures are taken during a hemodialysis treatment day and during a non-dialysis day. Interrater reliability between two different observers will be also calculated

DETAILED DESCRIPTION:
Patients suffering from End Stage Renal Disease are commonly involved in haemodialysis treatment, which is the most common treatment at this stage. Haemodialysis substitutes the renal function but is associated with several alterations that lead to decrease in functional capacity. Many studies show that functional capacity is significantly worse than their healthy sedentary age - matched counterparts. The purpose of the present study is to calculate values of absolute and relative intrarater reliability (dialysis vs non dialysis day) and interrater reliability of different physical function measures (Short Physical Performance Battery, one-leg balance, Timed Up and go, sit to stand to sit tests, triceps and handgrip strength, six-minute walking test).

ELIGIBILITY:
Inclusion Criteria:

* At least 3 months in hemodialysis treatment
* Clinically stable

Exclusion Criteria:

* Recent cardiac events (less than 3 months)
* Unable to exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with Chronic Kidney Diseases undergoing hemodialysis treatment
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline Short Physical Performance Battery at one week | It will perform the test three times with one week interval between the testing sessions, one before hemodialysis, and the other one next week during a non-dialysis day
  Assess lower extremity, which includes objective performance-based measure of balance (side-by-side, semitandem and tandem), endurance (4m gait speed) and strength (five chair stands). Each component was scored from 0 to 4 and when summed yielded SPPB scores between 0 (poor) and 12 (best).

SECONDARY OUTCOMES:
Change from baseline Gait speed at one week at one week | It will perform the test three times with one week interval between the testing sessions, one before hemodialysis, and the other one next week during a non-dialysis day
  Speed to cover 4 meters, in meters/second
Change from baseline One-leg standing test at one week | It will perform the test three times with one week interval between the testing sessions, one before hemodialysis, and the other one next week during a non-dialysis day
  Time achieved while standing on one leg
Change from baseline Timed up and go at one week | It will perform the test three times with one week interval between the testing sessions, one before hemodialysis, and the other one next week during a non-dialysis day
  Time to stand up, walk 3 meters, come back and sit down again
Change from baseline Sit to stand 10 test at one week | It will perform the test three times with one week interval between the testing sessions, one before hemodialysis, and the other one next week during a non-dialysis day
  Time to perform 10 repetitions sit to stand
Change from baseline Sit to stand 60 test at one week | It will perform the test three times with one week interval between the testing sessions, one before hemodialysis, and the other one next week during a non-dialysis day
  Sit to stand repetitions performed in 60 seconds
Change from baseline One-leg heel rise test at one week | It will perform the test three times with one week interval between the testing sessions, one before hemodialysis, and the other one next week during a non-dialysis day
  Number of heel rise repetitions achieved
Change from baseline 6 minutes walk test at one week | It will perform the test three times with one week interval between the testing sessions, one before hemodialysis, and the other one next week during a non-dialysis day
  Number of meters walked in 6 minutes
Change from baseline Handgrip at one week | It will perform the test three times with one week interval between the testing sessions, one before hemodialysis, and the other one next week during a non-dialysis day
  Bilateral handgrip strength

CONTACTS AND LOCATIONS:
Overall Officials: Vicent Esteve-Simó, PhD, Study Chair — Hospital de Terrassa
Locations (1):
- Hospital de Terrassa, Terrassa, Barcelona, Spain

REFERENCES:
- [Background] Esteve Simo V, Junque Jimenez A, Moreno Guzman F, Carneiro Oliveira J, Fulquet Nicolas M, Pou Potau M, Saurina Sole A, Duarte Gallego V, Tapia Gonzalez I, Ramirez de Arellano M. Benefits of a low intensity exercise programme during haemodialysis sessions in elderly patients. Nefrologia. 2015;35(4):385-94. doi: 10.1016/j.nefro.2015.03.006. Epub 2015 Jul 21. English, Spanish. PMID 26306966
- [Background] Segura-Orti E, Martinez-Olmos FJ. Test-retest reliability and minimal detectable change scores for sit-to-stand-to-sit tests, the six-minute walk test, the one-leg heel-rise test, and handgrip strength in people undergoing hemodialysis. Phys Ther. 2011 Aug;91(8):1244-52. doi: 10.2522/ptj.20100141. Epub 2011 Jun 30. PMID 21719637
- [Background] Ortega-Perez de Villar L, Martinez-Olmos FJ, Junque-Jimenez A, Amer-Cuenca JJ, Martinez-Gramage J, Mercer T, Segura-Orti E. Test-retest reliability and minimal detectable change scores for the short physical performance battery, one-legged standing test and timed up and go test in patients undergoing hemodialysis. PLoS One. 2018 Aug 22;13(8):e0201035. doi: 10.1371/journal.pone.0201035. eCollection 2018. PMID 30133445